CLINICAL TRIAL: NCT03549741
Title: Cabergoline As An Adjuvant To Clomiphene Citrate For Management Of Unexplained Infertility: Randomized Controlled Trial
Brief Title: Cabergoline As An Adjuvant To Clomiphene Citrate For Management Of Unexplained Infertility
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdeltawab Mhanny, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CabCC
Record Dates: First submitted 2018-05-26; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Cabergoline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): will receive a dose of Clomiphene citrate 50 mg tablet , 1 tab twice daily for 5 days from the third day of menses to the seven day and cabergoline 0.25 mg (half tablet) every 3 days (one package) first three months then Clomiphene citrate 50 mg tablet , 2 tabs twice daily for 5 days from the third day of menses to the seven day and cabergoline 0.25 mg (half tablet) every 3 days (one package)
  Interventions: Drug: Clomiphene Citrate 50mg; Drug: Cabergoline Oral Tablet
- control group (Active Comparator): will receive a dose of Clomiphene citrate and placebo tablets with same dose and duration
  Interventions: Drug: Clomiphene Citrate 50mg; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Clomiphene Citrate 50mg — oral tablets
Drug: Cabergoline Oral Tablet — oral tablets
  Arms: study group
Drug: Placebo Oral Tablet — oral tablets
  Arms: control group

SUMMARY:
Infertility refers to an inability to conceive after having regular unprotected sex. Infertility can also refer to the biological inability of an individual to contribute to conception, or to a female who cannot carry a pregnancy to full term. In many countries infertility refers to a couple that has failed to conceive after 12 months of regular sexual intercourse

ELIGIBILITY:
Inclusion Criteria:

* unexplained infertility, Primary or secondary.
* Absence of galactorrhoea.
* Normal serum prolactin.
* Normal hysterosalpingography.
* Normal spermogram.

Exclusion Criteria:

* Women on other line of treatment as aromatase inhibitors,gonadotrophins, or tamoxifen.
* Known hypersensitivity for cabergoline or clomiphene citrate.
* Other factors of infertility as tubal factor, uterine factor or male factor.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The number of mature follicles | 14 days
  the follicles reach the size of 18 mm